CLINICAL TRIAL: NCT06305260
Title: The LOTUS Trial: Lumbar Ultrasound Utility in Obstetric Patients With BMI > 40
Brief Title: LOTUS Trial: Lumbar Ultrasound in Obstetric Patients With BMI > 40
Acronym: LOTUS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00000324
Record Dates: First submitted 2023-12-11; First posted 2024-03-12 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Obesity, Morbid; Labor Pain
Keywords: Labor Epidural
MeSH Terms: conditions — Obesity, Morbid; Labor Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Lumbar Palpation (No Intervention): This group will include parturients who are randomized to traditional lumbar palpation prior to epidural placement. This is the current standard of care.
- Pre-procedural Lumbar Ultrasound (Experimental): This group will include parturients who are randomized to a pre-procedural lumbar ultrasound prior to epidural placement.
  Interventions: Diagnostic Test: Lumbar Ultrasound

INTERVENTIONS:
Diagnostic Test: Lumbar Ultrasound — Investigators will utilize our ultrasound machine to complete a pre-procedural lumbar ultrasound prior to epidural placement.
  Arms: Pre-procedural Lumbar Ultrasound

SUMMARY:
The goal of this clinical trial is to compare traditional palpation to pre-procedural lumbar ultrasound prior to epidural placement in obese (BMI >40) obstetric patient population. The main questions it aims to answer are:

* Is a pre-procedural lumbar ultrasound superior to traditional palpation in terms of total number of epidural needle redirections during epidural placement?
* Is there no difference in time to epidural loss between pre-procedural lumbar ultrasound and traditional palpation during epidural placement? Participants will be randomized to either a pre-procedural lumbar ultrasound or traditional palpation at the time of epidural placement.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* English Speaking
* BMI (Body Mass Index) > 40
* Ability to provide informed consent and verbally disclose their medical history

Exclusion Criteria:

* History of spine surgery, scoliosis, or other spinal abnormality which could complicate epidural placement
* Patients with platelet counts <70,000 or patients who are on anticoagulation, or patients who are on anticoagulation, both would exclude any patient from receiving an epidural.
* Minors
* Adults unable to make their own decisions or with cognitive issues or developmental delays
* Prisoners

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is only being completed in pregnant patients.
Enrollment: 150 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Epidural Redirects | Day of Epidural
  Total number of epidural needle redirections

SECONDARY OUTCOMES:
Total time to epidural space | Day of Epidural
  Total time to epidural space observed via loss of resistance.
Number of attempts at a different level | Day of Epidural
  Number of attempts at a different lumbar level.
Epidural replacement rate | Day of Epidural
  Includes epidurals that needed to be replaced because of failed epidural or inadequate pain relief
Patient satisfaction | 24 hours post-epidural
  Patient's satisfaction with epidural experience observed by a survey in post-partum

CONTACTS AND LOCATIONS:
Locations (1):
- MetroHealth Hospital, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided